CLINICAL TRIAL: NCT00991783
Title: A Clinical Trial to Evaluate the Effect of Fimasartan on Pharmacokinetics, and the Safety of Digoxin in Healthy Male Volunteers
Brief Title: A Study to Evaluate the Effect of Fimasartan on Pharmacokinetics, and the Safety of Digoxin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Choi, Director, Boryung Pharmaceutical Co., Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: A657-BR-CT-110
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-11

CONDITIONS: Essential Hypertension
Keywords: Fimasartan; Drug interaction
MeSH Terms: conditions — Essential Hypertension | interventions — Digoxin; fimasartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Digoxin + Fimasartan — Digoxin (7 days), Digoxin + Fimasartan (7 days)

SUMMARY:
The purpose of this study is to evaluate the effect of fimasartan on pharmacokinetics, and the safety of digoxin.

ELIGIBILITY:
Inclusion Criteria:

* age: 20 - 40 years
* sex: male
* body weight: greater than 55 kg
* written informed consent

Exclusion Criteria:

* known allergy to Fimasartan and digoxin
* existing cardiac or hematological diseases
* existing hepatic and renal diseases
* existing gastrointestinal diseases
* acute or chronic diseases which could affect drug absorption or metabolism history of any serious psychological disorder
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day 3 month ago
* participation in a clinical trial during the last 2 months prior to the start of the study

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
AUC, Cmax, Tmax, CL | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 15, 24 hours at 7 day and 28 day

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, Study Chair — Seoul National University Hospital